CLINICAL TRIAL: NCT05703100
Title: Relationship Between Lactate Profile and Fat Oxidation During Exercise
Brief Title: Lactate Profile and Fat Oxidation During Exercise
Acronym: LacFat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, Rocío Cupeiro, PhD, Physical Activity and Sports PhD (Associate Professor), Technical University of Madrid
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-061
Record Dates: First submitted 2023-01-11; First posted 2023-01-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Energy Metabolism
Keywords: lactate kinetics; exercise; energy metabolism; hyperthermia; glycogen depletion
MeSH Terms: conditions — Motor Activity; Hyperthermia | interventions — Diathermy

STUDY DESIGN:
Masking Description: No Masking is possible since participants and investigators know which type of test (control, hyperthermia and glycogen depletion) is being performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Maximal test on a cycle ergometer
  Interventions: Other: Incremental exercise test
- Hyperthermia (Experimental): Maximal test on a cycle ergometer at 35º-38º C room temperature
  Interventions: Other: Incremental exercise test under hyperthermia
- Glycogen depletion (Experimental): Maximal test on a cycle ergometer after a glycogen depletion protocol
  Interventions: Other: Incremental exercise test under glycogen depletion

INTERVENTIONS:
Other: Incremental exercise test — Maximal incremental exercise test on a cycle ergometer (5 min warm-up at 30W, and subsequent steps of 3 min with power increases of 30W)
  Other Names: Maximal incremental ergometry
  Arms: Control
Other: Incremental exercise test under hyperthermia — Maximal incremental exercise test on a cycle ergometer (5 min warm-up at 30W, and subsequent steps of 3 min with power increases of 30W) performed at a room temperature of 35-38ºC (degrees Celsius).
  Other Names: Maximal incremental ergometry with hyperthermia
  Arms: Hyperthermia
Other: Incremental exercise test under glycogen depletion — Maximal incremental exercise test on a cycle ergometer (5 min warm-up at 30W, and subsequent steps of 3 min with power increases of 30W) under glycogen depletion by performing an exercise protocol to deplete glycogen stores plus a low-carbohydrate diet 24 h before incremental testing
  Other Names: Maximal incremental ergometry with glycogen depletion
  Arms: Glycogen depletion

SUMMARY:
The goal of this clinical trial is to test whether changes in lactate kinetics during exercise (due to glycogen depletion or hyperthermia) alter the pattern of fat oxidation during a maximal incremental cycle ergometer test in healthy young active people. The main questions it aims to answer are:

* Will a rightward shift in lactate kinetics, induced by a previous glycogen depletion, produce a rightward shift in fat oxidation?
* Will a leftward shift in lactate kinetics due to an increase in ambient temperature produce a leftward shift in fat oxidation?

Participants will perform three maximal incremental tests in three different conditions:

* one in the control condition;
* one with glycogen depletion;
* and one with ambient heat (the latter two in randomized, counterbalanced order).

DETAILED DESCRIPTION:
Introduction Lactate has three major functions: it is an energy substrate, it is a gluconeogenic precursor, and it is a signalling molecule (1). Among the signalling functions is that of modulating skeletal muscle metabolism, as a regulator of fat oxidation at both the autocrine and paracrine levels. At the autocrine level, lactate increases the levels of Acetyl-coenzyme A (CoA) inside the mitochondria and, consequently, the levels of Malonyl-CoA. The increase in Malonyl-CoA concentration inhibits Carnitine PalmitoylTransferase 1 (CPT1), which is one of the transporters of fatty acids into the mitochondria (2). At the paracrine level, an increase in blood lactate concentration reduces the release of fatty acids into the blood by adipose tissue (3). This occurs because the G protein-coupled receptor present in adipose tissue inhibits the release of fatty acids into the blood when the blood lactate concentration increases (4). However, in vivo, only an inverse correlation between blood lactate concentration and fatty acid oxidation has been demonstrated (5,6). Therefore, the main objective of the study is to observe whether the pattern of fat oxidation during a maximal incremental cycle ergometer trial is altered due to changes in lactate kinetics during the given trial. For this purpose, three maximal trials will be performed with the same loading protocol (intensity and progression of the same), but different physiological conditions (normal vs. previous glycogen depletion vs. environmental hyperthermia).

Procedures Consent to participate (signature of informed consent) will be requested from all volunteers who meet the inclusion criteria.

The tests that will be performed throughout this study will be the following:

1. At the first appointment, you will be asked about your medical history. Then, if appropriate, an assessment of your body composition by dual X-ray absorptiometry (DEXA) will be performed,
2. In the second appointment, spirometry, an electrocardiogram at rest, and finally, an ergospirometric trial will be performed.
3. In the third, fourth, and fifth visits, three maximal exercise trials will be performed, one each day. Of the three maximum ergospirometric trials that will be performed, one will be in a hot environment -approximately 38º Celsius (ºC) ambient temperature- and the other in a state of glycogen depletion. A glycogen depletion protocol and a low-carbohydrate diet will be performed before the maximal ergospirometric trial in the glycogen-depleted state, while the other two trials (simple maximal trial and hot-environment maximal trial) will be performed after 24h of a high-carbohydrate diet.
4. The order of performance of each protocol will be randomized, provided that the glycogen depletion protocol is performed at the visit prior to the maximal ergospirometric trial under glycogen depletion. The depletion protocol consists of a 60-minute continuous cycle ergometer effort at the power associated with 60% of the maximal oxygen uptake (VO2) followed by six 30-second maximal efforts with four minutes of recovery. After this glycogen depletion exercise protocol, the participant will follow a low-carbohydrate diet (2% carbohydrate, 78% fat, and 20% protein), until the time of the ergospirometric trial under glycogen depletion status.

ELIGIBILITY:
Inclusion Criteria:

* Perform endurance training with a volume of between 3 and 12h/week
* In women, having regular menstrual cycles (25-35 days length)
* In women, being able to perform the test without menstrual discomfort or pain and without having taken anti-inflammatory or analgesic drugs

Exclusion Criteria:

* Suffering from any previous disease, disorder or ailment that could affect the results of the study variables
* Smoking
* In women, using any type of hormonal contraceptive
* In women, having heavy menstrual bleeding, detected with the menstrual bleeding questionnaire proposed by Wyatt et al. (2001)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Blood lactate concentration | Through study completion, an average of 5 months
  Lactate concentration, expressed in mMol/L (Millimoles Per Liter), measured in capillary blood using a lactate analyser. Lactate concentration is measured in the capillary blood extracted from the fingertip, during the tests performed in the different situations (control, glycogen depletion and hyperthermia)
Fat oxidation | Through study completion, an average of 5 months
  Fat oxidation, expressed in g/min, is indirectly measured through the analysis of the gas composition of breathing (O2 and CO2), using a gas analyser. Fat oxidation is measured during the tests performed in the different situations (control, glycogen depletion and hyperthermia)

SECONDARY OUTCOMES:
Heart Rate | Through study completion, an average of 5 months
  Heart rate, expressed in bpm (beats per minute), is measured using a pulsometer. Heart rate is measured during the tests performed in the different situations (control, glycogen depletion and hyperthermia)
Power output | Through study completion, an average of 5 months
  Power output, expressed in watts, is measured with a cycle ergometer. Power output is measured during the tests performed in the different situations (control, glycogen depletion and hyperthermia)

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Cupeiro, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Laboratorio de Fisiología del Esfuerzo. Facultad de Ciencias de la Actividad Física y del Deporte (INEF), Madrid, Spain

REFERENCES:
- [Background] Wyatt KM, Dimmock PW, Walker TJ, O'Brien PM. Determination of total menstrual blood loss. Fertil Steril. 2001 Jul;76(1):125-31. doi: 10.1016/s0015-0282(01)01847-7. PMID 11438330
- [Derived] Benitez-Munoz JA, Guisado-Cuadrado I, Rojo-Tirado M, Alcocer-Ayuga M, Romero-Parra N, Peinado AB, Cupeiro R. Females have better metabolic flexibility in different metabolically challenging stimuli. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-12. doi: 10.1139/apnm-2024-0217. Epub 2024 Oct 22. PMID 39437435